CLINICAL TRIAL: NCT07174713
Title: REverse LuNg Airway and Vascular RemOdeling in Asthma ReMission (ReNORM)
Acronym: ReNORM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Grace Parraga, Principal Investigator, Western University, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROB0061
Record Dates: First submitted 2025-08-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Asthma; Eosinophilic
Keywords: Hyperpolarized Xenon MRI; Clinical Remission; Biologic Therapy; Airway Remodeling
MeSH Terms: conditions — Pulmonary Eosinophilia; Airway Remodeling | interventions — Biological Therapy

STUDY DESIGN:
Intervention Model Description: Parallel assignment of participants to one of two arms: (1) patients with severe asthma initiating biologic therapy, and (2) healthy volunteers serving as controls. Asthma patients are followed over 2 years to assess clinical, imaging, and histologic responses to biologic treatment. A randomized subset of asthma participants undergoes MRI-guided bronchoscopy to correlate imaging with histopathology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma - Biologic Therapy (Experimental): Participants with severe asthma (GINA 5) who are eligible to begin biologic therapy. Participants will undergo serial assessment with pulmonary imaging (CT, MRI), lung function testing, sputum collection, and symptom questionnaires. A subset of participants (~15%) will be randomized to undergo MRI-guided bronchoscopy with airway sampling at baseline and 2 years.
  Interventions: Biological: Biologic Therapy
- Healthy Control (No Intervention): Age- and sex-matched healthy participants with no history of lung disease. Participants will undergo pulmonary imaging (CT, MRI) and lung function testing at baseline and follow-up for comparison with the asthma group. No therapeutic intervention will be provided.

INTERVENTIONS:
Biological: Biologic Therapy — Participants with severe asthma (GINA 5) who are eligible to begin biologic therapy. Participants will undergo serial assessment with pulmonary imaging (CT, MRI), lung function testing, sputum collection, and symptom questionnaires. A subset of participants (~15%) will be randomized to undergo MRI-guided bronchoscopy with airway sampling at baseline and 2 years.
  Arms: Asthma - Biologic Therapy

SUMMARY:
In this program of research, the investigators aim to answer the question: In patients with asthma aged 18-80, how do the lung airways and vessels respond to biologic therapy and what role does age and asthma duration have in this response? While about 4.6 million Canadians live with asthma, ~5-10% of patients have severe asthma meaning that multiple inhaled and systemic oral corticosteroid treatments have failed to improve symptoms and exacerbations, leading to lost work and school days and substantially diminished ability to participate in normal life. For such people, the vast majority of whom are middle aged and remember asthma as part of their entire lifespan, biologic immunomodulator therapies, which block the function of asthma inflammatory pathways, provide a final step-up therapy option. There is emerging evidence that prescribed in the right patient at the right time, the right biologic can result in clinical remission of asthma. While spontaneous clinical remission of asthma is rare, it has been documented in children in whom lung growth and remodeling is still possible. It remains unknown whether clinical remission in adults is accompanied by the reversal of pathologic remodeling, at the level of the airways and pulmonary vessels. This is critical to elucidate as investigators and physicians move forward with currently proposed criteria for "complete asthma remission". The inconvenient truth about asthma and age is that in older adult lungs, exposed to years of infection, exacerbations, smooth muscle remodeling and pulmonary vascular shunt, the mechanisms by which complete pathologic remission may be achieved are complex and poorly understood.

To address this knowledge gap, the investigators will evaluate 150 patients (Vancouver, Ottawa, Hamilton, London) (in three age tertiles 18-29; 30-59; 60-80) with severe asthma and 50 age- and sex matched healthy volunteers over 2-years using chest CT, MRI and pulmonary function tests. The investigators will use the pulmonary imaging measurements to generate an imaging-index of normal airway structure and function which will be compared with and significantly correlate with MR-guided bronchoscopic sample measurements made before and after 1-/2-years of treatment. The investigators will reveal the pathobiologic relationship between age, asthma duration, clinical remission and imaging normalization with direct comparison to histology-based airway measurements.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must meet all the following criteria:

1. Participant understands study procedures and is willing to participate in the study as indicated by the patient's signature.
2. Provision of written, informed consent prior to any study specific procedures.
3. Males and females aged 18 to 80 years.
4. Either diagnosed with severe asthma (GINA Step 5) and newly eligible for biologic therapy (based on ACQ-5, current treatment, exacerbation history, and blood eosinophils in accordance with approved criteria for omalizumab, mepolizumab, benralizumab, dupilumab, or tezepelumab), or a healthy volunteer with no history of chronic lung disease, matched by age and sex. Healthy participants must have a lifetime combustible tobacco and/or cannabis (including vaping) consumption of ≤5 pack-years.
5. Women of childbearing potential (after menarche) must ensure that they are using an effective form of birth control for at least 2 months prior to each imaging visit. Examples of effective birth control include:

   1. True sexual abstinence
   2. A vasectomized sexual partner
   3. Implanon®
   4. Female sterilization by tubal occlusion
   5. Effective intrauterine device (IUD)/levonogestrel intrauterine system (IUS)
   6. Depo-Provera™ injections
   7. Oral contraceptive
   8. Evra Patch™
   9. Nuvaring™
6. Women of childbearing potential (after menarche) must agree to use a highly effective form of birth control, as defined above, from enrollment, throughout the study duration, and 8 weeks after last dose of study drug, with negative urine pregnancy test result at Visit 1-5.
7. Male participants who are sexually active must agree to use a double barrier method of contraception (male condom with diaphragm or male condom with cervical cap) from the first dose of the study drug until 8 weeks after last dose

Exclusion Criteria:

Participants fulfilling any of the following criteria are not eligible for inclusion in this study:

1. Patient has an implanted mechanically, electrically, or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist).
2. In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI or CT, such as severe claustrophobia.
3. Participants who are pregnant, breastfeeding or have a positive pregnancy test at initial screening visit.
4. Participant is unable to perform spirometry or plethysmography maneuvers.
5. Participant is unable to perform MRI and CT breath-hold maneuvers.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Determine extent of imaging-based remission in patients with severe asthma following 1 and 2 years of biologic therapy | from baseline to year 1 and year 2
  Measured using 129Xe ventilation defect percent (VDP)
Measure the extent and timing of clinical remission in patients with severe asthma as measured by changes in spirometry measurements of FEV1 and FVC | from baseline to 1 year and 2 years
  Measured using forced expiratory volume in 1 second and forced vital capacity
To determine the extent and timing of clinical remission in patients with severe asthma using symptoms scores of ACQ-5 and ACT | From baseline to 1 year and 2 years
  Measured using changes in asthma control questionnaire and asthma control test
Determine the extent and timing of imaging-based remission in patients with severe asthma using CT airway and vessel morphology | From baseline to 1 year and 2 years
  Measured using computed tomography (CT) airway and vessel metrics
To determine the extent and timing of clinical remission using the clinical outcome of frequency of asthma exacerbations in patients with severe asthma | from baseline to 1 year and 2 years
  Measured using the number of asthma exacerbations
To determine the extent and timing of clinical remission of patients with severe asthma using the clinical outcome of OCS use | From baseline to 1 year and 2 years
  Measured by the frequency of oral corticosteroid usage
Determine the extent and timing of clinical remission in patients with severe asthma as measured by sputum and blood eosinophil counts | From baseline to 1 year and 2 years
  Measured using blood and sputum eosinophil counts

SECONDARY OUTCOMES:
Timing and proportion of patients achieving clinical remission after biologic treatment as measured by FEV1 and FVC. | From baseline to 1 year and 2 years
  Measured using forced expiratory volume at 1 second and forced vital capacity.
To determine the timing and proportion of patients achieving clinical remission as measured by ACQ-5 and ACT questionnaires. | From baseline to 1 year and 2 years
  Measured by asthma control questionnaire and asthma control test questionnaire scores.
Determine the timing and proportion of patients with severe asthma achieving clinical remission after biologic treatment using FeNO. | From baseline to 1 year and 2 years
  Measured using fractional exhaled nitric oxide (FeNO)
Determine the timing and proportion of patients with severe asthma achieving clinical remission using DLco. | From baseline to 1 year and 2 years
  Measured using diffusing capacity of the lung for carbon monoxide (DLco)
Determine the timing and proportion of patients with severe asthma achieving clinical remission after biologic treatment using SGRQ score. | From baseline to 1 year and 2 years.
  Measured using St. George's Respiratory Questionnaire (SGRQ) score.
Determine the timing and proportion of patients with severe asthma achieving clinical remission on biologic treatment using AQLQ scores. | From baseline to 1 year and 2 years
  Measured using the Asthma Quality of Life Questionnaire (AQLQ) score.
Determine the timing and proportion of patients with severe asthma achieving imaging normalization after biologic treatment using 129-Xe MRI VDP | From baseline to 1 year and 2 years
  Measured using the changes in 129-xenon MRI ventilation defect percent (VDP)
Determine the timing and proportion of patients with severe asthma achieving imaging normalization after biologic treatment using CT metrics | From baseline to 1 year and 2 years
  Measured using computed tomography (CT) mucus-score, airway dimensions and vascular pruning
Determine the timing and proportion of patients with severe asthma achieving imaging normalization after biologic treatment using DLco. | From baseline to 1 year and 2 years
  Measured using diffusing capacity of the lung for carbon monoxide (DLco)
Determine the timing and proportion of patients with severe asthma achieving imaging normalization after biologic treatment using RV/TLC | From baseline to 1 year and 2 years
  Measured using the ratio of residual volume to total lung capacity (RV/TLC)
Determine the timing and proportion of patients with severe asthma achieving imaging normalization after biologic treatment using FRC. | From baseline to 1 year and 2 years
  Measured using functional residual capacity (FRC).
Determine the relationships between clinical and imaging remission and generate predictive models for their achievement using changes in VDP | from baseline to 12-weeks and 2-years
  Measured using ventilation defect percent (VDP)
Determine the relationship between clinical and imaging remission and generate predictive models for their achievement using changes in CT. | From baseline to 12-weeks and 2-years
  Measured using computed tomography (CT) airway wall thickness, mucus metrics
Determine the relationships between clinical and imaging remission and generate predictive models for their achievement using FeNO. | From baseline to 12-weeks and 2-years
  Measured using forced exhaled nitric oxide (FeNO).
Determine the relationships between clinical and imaging remission and generate predictive models for their achievement using ACQ-5 and ACT scores. | From baseline to 12-weeks and 2-years.
  Measured using asthma control questionnaire and asthma control test scores.
Determine the relationships between clinical and imaging remission and generate predictive models for their achievement using sputum biomarkers. | From baseline to 12-weeks and 2-years
  Measured using sputum eosinophil and cell count values
Determine the relationships between clinical and imaging remission and generate predictive models for their achievement using exacerbation history. | From baseline to 12-weeks and 2-years.
  Measured using patient's reported exacerbation history.

OTHER OUTCOMES:
Quantify the relationships of imaging and pathologic markers of remodeling and develop a non-invasive imaging-index lung normalization. | From baseline (Day 0) to year 2
  Measured using bronchoscopic airway histology (epithelial thickness, smooth muscle mass, vascularity).
Quantify the relationships of imaging and pathologic markers of remodeling and develop a non-invasive imaging-index lung normalization using MRI/CT correlations with histologic changes | From baseline to 2 years.
  Measured using MRI, CT and histology values
Quantify the relationships of imaging and pathologic markers of remodeling and develop a non-invasive imaging-index lung normalization using MRI/CT fusion data | From baseline to 2 years.
  Measured using MRI and CT measurements

CONTACTS AND LOCATIONS:
Overall Officials: Grace Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No